CLINICAL TRIAL: NCT00003696
Title: Phase III Study of Cyclophosphamide, Doxorubicin and Etoposide Compared to Carboplatin and Taxol in Patients With Extensive Disease Small Cell Lung Cancer
Brief Title: Combination Chemotherapy in Treating Patients Who Have Extensive-Stage Small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Commissie Voor Klinisch Toegepast Onderzoek (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066803; CKVO-9802; DUT-KWF-CKVO-9802; EU-98059
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2001-11

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Carboplatin; Cyclophosphamide; Doxorubicin; Etoposide; Paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which combination chemotherapy regimen is most effective for extensive-stage small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of two combination chemotherapy regimens in treating patients with extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effect of cyclophosphamide, doxorubicin, and etoposide with carboplatin and paclitaxel on progression free survival in patients with extensive stage small cell lung cancer.
* Compare the overall survival, response rate, duration of response, and toxic effects of these regimens in these patients.

OUTLINE: This is a randomized study. Patients are stratified according to institute and performance status (0-1 vs 2-3).

Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive cyclophosphamide IV and doxorubicin IV on day 1, and etoposide IV on days 1-3 every 3 weeks.
* Arm II: Patients receive carboplatin IV followed by paclitaxel IV over 3 hours on day 1 every 3 weeks.

Patients with stable or responding disease are treated for up to 5 courses.

Patients are followed every 4 weeks.

PROJECTED ACCRUAL: A total of 250 patients (125 per treatment arm) will be accrued within 24 months for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven extensive stage small cell lung cancer, not previously treated with chemotherapy or radiotherapy except for symptomatic brain metastases
* Measurable or evaluable disease

  * Ascites, pleural effusions, osteolytic and osteoblastic bone metastases are not measurable or evaluable

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-3

Life expectancy:

* Not specified

Hematopoietic:

* Platelet count at least 100,000/mm^3
* Absolute neutrophil count at least 2,000/mm^3

Hepatic:

* Bilirubin no greater than 1.25 times upper limit of normal (unless due to liver metastases)

Renal:

* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No cardiac failure or rhythm disturbances requiring medication

Other:

* No history of hypersensitivity to castor oil
* No active uncontrolled infection
* No nonmalignant disease presenting a poor medical risk
* Not pregnant
* Fertile patients must use effective contraception during and for 3 months after the study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy

Chemotherapy:

* See Disease Characteristics
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy

Radiotherapy:

* See Disease Characteristics
* Palliative radiotherapy allowed (indicator lesion should be outside of irradiated field)

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 1998-10

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Overall survival
Response rate
Duration of response
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Egbert F. Smit, MD, Study Chair — Free University Medical Center
Locations (1):
- Vrije Universiteit Medisch Centrum, Amsterdam, Netherlands